CLINICAL TRIAL: NCT06863103
Title: Dentists' Experiences From Treating Children With Extensive Dental Treatment Needs
Brief Title: Treating Children With Extensive Dental Needs
Status: Enrolling by invitation | Type: Observational
Sponsor: Malmö University (Other)
Responsible Party: Sponsor
Other Study IDs: MAU 2024/122
Record Dates: First submitted 2024-12-05; First posted 2025-03-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Dental Caries; Tooth Extraction; Conscious Sedation; Attitude; Anesthesia, General
Keywords: grounded theory; dentist; pediatric dentistry; dental caries; ethical stress
MeSH Terms: conditions — Dental Caries; Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Child-treating dentists: Dentists meeting young children with extensive treatment need

SUMMARY:
The goal of this qualitative study, using Grounded Theory, is to gain deeper knowledge about dentists' experiences from treating in particular young children with an extensive treatment need (mainly due to caries).

The main question is to find out more about the dentists' reactions, feelings, perceived stress, and thoughts in general when meeting and treating young children with many carious lesions. The investigators also want to gain better understanding of how dentists think about reporting children who might be subject for maltreatment.

DETAILED DESCRIPTION:
BACKGROUND: Severe or extensive caries is a condition that affects a large number of children yearly. This could lead to serious consequences for the affected child such as pain, many dental visits, risk for poorer oral health, and poor esthetics. In many cases, there is a connection to lack of care, whereby dental professionals has an obligation to file a report to social services regarding concerns of maltreatment.

The dental care includes a wide spectrum of measures, from information och oral health preventive actions, to filling therapies and tooth extractions. I many cases the disease is so extensive that the child needs to be referred to a pediatric dentistry specialist clinic in order to get treatment under sedation or general anesthesia. This is more prevalent the younger the child is. Dental treatments performed under general anesthesia or sedation is often more radical and tooth extraction is a common therapy for teeth with extensive decay.

As a dentist, in charge of initial care and treatment, taking care of children who might not know or understand why they have to undergo treatment, or that maybe are scared or suffer from pain, might affect the general wellbeing of the dentist. Perception of stress, especially ethical stress, can further affect how dentists make treatment decisions, among other things. Despite this, the knowledge of how dentists perceive and are affected by meeting and treating children with extensive need for dental care, is unsatisfactory.

RESEARCH QUESTION How do dentists experience meeting and treating children with an extensive need for dental care? How is extensive need for dental care looked upon in relation to potential report to social services?

METHODS AND INFORMANTS This project will use Grounded Theory, that is a qualitative research method. When knowledge and theories are lacking within a certain area, common hypotheses testing methods are less suitable. Instead, by using qualitative research methods, information can be collected from individuals with experience from the area of interest. Some methods, like Grounded Theory, can lead to results that might form a base for formulating hypothesis that later can be tested in studies using quantitative/hypotheses testing methods.

In this project, interviews will be held with dentists (informants) that work within public dental care, and specialised dental care, i.e. specialists in pediatric dentistry. During the interviews a so called thematic interview guide with open themes is used, rather than using semi-structured that might lead what the informants choose to talk about. Intended themes in the interview guide concerns the following: experiences of treating children with extensive need for treatment, reflections upon reporting to social services, experiences of child patients reactions and abilities to handle dental treatment, thoughts about legal guardians being present in the operating room, experiences of different coping strategies, or anything else that the informant brings to the table. Informants will be general dental practitioners working with child dental care, mainly from county of Scania, and specialist in pediatric dentistry or post-graduate students becoming such specialists. The specialist cohort is recruited from all over Sweden.

The investigators plan to interview up to 25 dentists. The informants will be recruited to include different experiences, and backgrounds, e.g. different ages, years as dentist, general dental practitioner or specialist, public dental clinic or private clinic, working in city or rural area.

The interviews will take approximately one hour and will be recorded digitally, and the interviews can be performed both digitally or in a direct meeting, but over telephone is also a possibility. The interviews will be transcribed verbatim and analyzed according to preset routines according to to the chosen method, Grounded Theory. Interviews and analyses takes place parallell. The transcribed interviews will be analyzed, and through these analyses so called categories emerges, that describes what the experiences are about. These codes will then be merged into preliminary categories. In the following axial coding process, the preliminary categories will be further developed by identifying dimensions and characteristics, leading up to sub-categories. Relations data and categories is sought for, thus creating a "new whole". Selective coding will lead to data saturation and validation. The former can also be achieved by re-code already retreived data. In the results, there is also a core category that can be described as the most central and crucial aspects of the research questions being studied.

it is not applicable to calculate sample size when using qualitative method such as Grounded Theory. Instead, participants will be included until saturation in data is achieved, meaning that new information can not any longer be obtained.

KNOWLEDGE GAINS Grounded Theory is a theory generating method, especially suitable for research areas where existing theories are scarce or totally lacking. Today, a lot of research within medical and dental fields takes the investigator's perspective. It is highly crucial that also the directly affected are involved, i.e. the patients.

ELIGIBILITY:
Inclusion Criteria:

* Dentists, both general dental practitioners and specialist, or those under training to become specialist in pediatric dentistry.

Exclusion Criteria:

-

Max Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Dentists, both general dental practitioners and specialist, or those under training to become specialist in pediatric dentistry.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-03-26 (Actual); Primary Completion 2025-12-25 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Dentists' attitudes on handling children with extensive treatment need | The data will be collected and analyzed over a period of 12 months.
  This study aims to identify and categorize the main themes that emerge from qualitative interviews with dentists who treat children with extensive dental needs. The themes will be derived using grounded theory methodology, focusing on the challenges, strategies, and outcomes associated with providing care to this patient population. By analyzing data, codes will be identified, leading up to conceptual categories that in the end will form a core-category, a new theory.

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Berlin, PhD, Principal Investigator — Malmö University, Faculty of Odontology
Locations (1):
- Faculty of Odontology, Malmo University, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared.

REFERENCES:
- [Background] Kassebaum NJ, Bernabe E, Dahiya M, Bhandari B, Murray CJ, Marcenes W. Global burden of untreated caries: a systematic review and metaregression. J Dent Res. 2015 May;94(5):650-8. doi: 10.1177/0022034515573272. Epub 2015 Mar 4. PMID 25740856
- [Background] Griffen AL, Schneiderman LJ. Ethical issues in managing the noncompliant child. Pediatr Dent. 1992 May-Jun;14(3):178-83. PMID 1528787
- [Background] Farokh-Gisour E, Hatamvand M. Investigation of Stress Level Among Dentistry Students, General Dentists, and Pediatric Dental Specialists During Performing Pediatric Dentistry in Kerman, Iran, in 2017. Open Dent J. 2018 Sep 28;12:631-637. doi: 10.2174/1745017901814010631. eCollection 2018. PMID 30369972
- [Background] "Dellve L, Henning Abrahamsson K, Trulsson U, Hallberg LR-M. Grounded theory in public health research. In: Hallberg LR-M, ed. Qualitative methods in public health research: theoretical foundations and practical examples. Lund: Studentlitteratur, 2002; 137-173."
- [Background] Kvist T, Wickstrom A, Miglis I, Dahllof G. The dilemma of reporting suspicions of child maltreatment in pediatric dentistry. Eur J Oral Sci. 2014 Oct;122(5):332-8. doi: 10.1111/eos.12143. Epub 2014 Jul 11. PMID 25039643
- [Background] Kizilci E, Kizilay F, Mahyaddinova T, Muhtaroglu S, Kolcakoglu K. Stress levels of a group of dentists while providing dental care under clinical, deep sedation, and general anesthesia. Clin Oral Investig. 2023 Jul;27(7):3601-3609. doi: 10.1007/s00784-023-04973-9. Epub 2023 Mar 30. PMID 36995430
- [Background] Glaser B, Strauss A. The discovery of grounded theory: strategies for qualitative research. New York: Aldine de Gruyter, 1967.
- [Result] Davidovich E, Pessov Y, Baniel A, Ram D. Levels of Stress among General Practitioners, Students and Specialists In Pediatric Dentistry during Dental Treatment. J Clin Pediatr Dent. 2015 Fall;39(5):419-22. doi: 10.17796/1053-4628-39.5.419. PMID 26551363